CLINICAL TRIAL: NCT06759116
Title: Analgesic Effect of Fentanyl Vs Dexmedetomidine As Adjuvant to Bupivacaine in Combined IPACK and Adductor Canal Block After Knee Surgeries
Brief Title: Comparison Between Fentanyl and Dexmedetomidine As Adjuvant to Bupivacaine in Combined IPACK and Adductor Canal Block for Postoperative Analgesia After Knee Surgeries
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Dina Abdelhameed Elsadek Salem, principle investigator, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 940
Record Dates: First submitted 2024-12-29; First posted 2025-01-06 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-12

CONDITIONS: Analgesia, Postoperative
Keywords: fentanyl; dexamedetomidine; analgesia; IPACK and adductor canal block; knee surgeries
MeSH Terms: conditions — Agnosia | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Analgesic Effect of Fentanyl versus Dexmedetomidine as Adjuvants to Bupivacaine in combined IPACK and Adductor Canal Block after Knee Surgeries
Who Masked: Participant, Outcomes Assessor
Masking Description: anesthetist not sharing in the study will assess patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (group C) (Active Comparator): The patient receive unilateral ultrasound guided combined IPACK and ACB with bupivacaine only. two syringes , one for each block , each one contains (20 mL of 0.25% bupivacaine and 1 ml saline)
  Interventions: Procedure: Control group
- Fentanyl group (group F) (Active Comparator): The patient receive unilateral ultrasound guided combined IPACK and ACB with bupivacaine only. two syringes , one for each block , each one contains (20 mL of 0.25% bupivacaine and 50 mcg fentanyl)
  Interventions: Procedure: Fentanyl group
- Dexmedetomidine group (group D) (Active Comparator): The patient receive unilateral ultrasound guided combined IPACK and ACB with bupivacaine only. two syringes , one for each block , each one contains (20 mL of 0.25% bupivacaine and 1 ug/kg dexmedetomidine not exceeding 100 ug (to be completed to 1mL with normal saline if needed). )
  Interventions: Procedure: Dexmedetomidine group

INTERVENTIONS:
Procedure: Control group — The patient receive unilateral ultrasound guided combined IPACK and ACB with bupivacaine only. two syringes , one for each block , each one contains (20 mL of 0.25% bupivacaine and 1 ml saline)
  Arms: Control group (group C)
Procedure: Fentanyl group — The patient receive unilateral ultrasound guided combined IPACK and ACB with bupivacaine only. two syringes , one for each block , each one contains (20 mL of 0.25% bupivacaine and 50 mcg fentanyl)
  Arms: Fentanyl group (group F)
Procedure: Dexmedetomidine group — The patient receive unilateral ultrasound guided combined IPACK and ACB with bupivacaine only. two syringes , one for each block , each one contains (20 mL of 0.25% bupivacaine and 1 ug/kg dexmedetomidine not exceeding 100 ug (to be completed to 1mL with normal saline if needed). )
  Arms: Dexmedetomidine group (group D)

SUMMARY:
This study will be undertaken to compare the analgesic effects of of fentanyl versus dexmedetomidine as adjuvant to bupivacaine in combined IPACK and ACB for pain management after total knee arthroplasty.

DETAILED DESCRIPTION:
* To measure the total amount of rescue analgesic consumption in the first 48 hours post-operatively in each group
* To assess pain score in each group by using Numerical Rating Scale (NRS) at rest (static) and during flexion or extension of knee (dynamic) at different time points: PACU, 2 hrs, 4 hrs, 8 hrs, 12 hrs, 24 hrs and 48 hrs.
* To measure the time of first request of rescue analgesia in each group
* To record the incidence of adverse events (hematoma, local anesthetic toxicity, infection, nausea and vomiting) and length of hospital stay.
* Over all patients' satisfaction: The patients will be asked to rate the overall degree of satisfaction of the analgesia by using a 5-points Likert-like verbal scale (1 = very dissatisfied analgesia, 2 = dissatisfied analgesia, and 3 = neutral, 4=satisfied analgesia, and 5=very satisfied analgesia).

ELIGIBILITY:
Inclusion Criteria:

1 - Patient acceptance 2. Cooperative patients 3. Age: ≥21 and 85< years' old 4. Sex: both sexes (males or females). 5. Physical status: ASA Ι & II& Ш. 6. Body Mass Index (BMI): ≤ 35 kg/m2. 7. Type of operation: elective unilateral knee surgeries (TKA, ACL, knee arthroscopy)

Exclusion Criteria:

. Patient with any contraindications of regional blocks (as coagulopathy or local infection at injection site) 2. Patients with known history of allergy to the study drugs (bupivacaine, dexmedetomidine and fentanyl).

3. Advanced hepatic, renal, cardiovascular, neurologic and respiratory diseases.

4.Chronic opioid use (more than 3 months or daily oral morphine > 5 mg /day for 1 month)

-

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-07-10 (Estimated); Study Completion 2025-08-10 (Estimated)

PRIMARY OUTCOMES:
● The total amount of rescue analgesic consumption (tramadol) | For 48 hrs
  ● The total amount of rescue analgesic consumption (tramadol) postoperatively in each group
Pain intensity by using Numerical Rating Scale (NRS) at rest (static) and during flexion or extension of knee (dynamic) at different time points | 0 hours (basal) ( on arrival to PACU), 2 hrs, 4 hrs, 8 hrs, 12 hrs, 24 hrs and 48 hrs
  NRS is 10 cm line numbered from 0 to 10, patients instructed to circle the number that represents his/her pain intensity (0=no pain and 10=maximum pain)

SECONDARY OUTCOMES:
The time to first request of rescue analgesia (tramadol) | 24 hours postoperative
  The time to first request of rescue analgesia (tramadol) (time from end of local anesthetics injection till time of NRS ≥ 3)
The length of hospital stays | For 48-72 hrs
  The length of hospital stays (number of hospital stay days starting from discharge from PACU till discharge home).
The incidence of adverse events | For 48 hrs
  The incidence of adverse events (hematoma, local anesthetic toxicity, infection, nausea and vomiting).
patient's satisfaction | For 48 hrs
  patient's satisfaction: The patients will be asked to rate the overall degree of satisfaction of the analgesia by using a 5-points Likert-like verbal scale (1 = very dissatisfied analgesia, 2 = dissatisfied analgesia, and 3 = neutral, 4=satisfied analgesia, and 5=very satisfied analgesia)

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of human medicine, Zagazig university hospitals, El Sharkia, Egypt

IPD SHARING:
Plan to Share IPD: No